CLINICAL TRIAL: NCT00607893
Title: Oxidative Stress in Sleep Apnea and Cardiac Disease
Brief Title: Efficacy of Continuous Positive Airway Pressure in Reducing Oxidative Stress in Individuals With Sleep Apnea
Acronym: SASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Reena Mehra, Associate Professor, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 562; K23HL079114 (NIH)
Record Dates: First submitted 2008-01-25; First posted 2008-02-06 (Estimated); Results first posted 2017-09-15 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-08

CONDITIONS: Sleep Apnea Syndromes; Oxidative Stress; Cardiovascular Diseases
Keywords: Sleep-Disordered Breathing
MeSH Terms: conditions — Sleep Apnea Syndromes; Cardiovascular Diseases | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham CPAP (Sham Comparator): Participants will receive sham continuous positive airway pressure (CPAP) for a 2 month period. Sham CPAP involves wearing a device that appears similar to a standard CPAP device, but administers a negligible pressure. Adherence will be tracked while the participant wears the device.
  Interventions: Device: Sham CPAP
- Treatment CPAP (Active Comparator): Participants will receive continuous positive airway pressure for a 2 month period. The optimal treatment pressure will be identified during a titration study prior to trial enrollment. Adherence will be tracked while the participant wears the device.
  Interventions: Device: Continuous Positive Airway Pressure (CPAP)

INTERVENTIONS:
Device: Continuous Positive Airway Pressure (CPAP) — Participants will use the higher pressure CPAP, as determined by an in-laboratory attended titration study, every night for 12 weeks.
  Arms: Treatment CPAP
Device: Sham CPAP — Participants will use the lower pressure CPAP every night for 8 weeks.
  Arms: Sham CPAP

SUMMARY:
Sleep-disordered breathing (SDB) is a condition in which a person experiences frequent breathing pauses during sleep, also known as sleep apnea. There is evidence that the recurrent sleep arousal and associated shortage of oxygen in the body may increase risk for cardiovascular disease (CVD). It is believed that treatment with continuous positive airway pressure (CPAP) may reduce certain risk factors for heart disease, including markers of inflammation and oxidative stress. This study will evaluate the effectiveness of CPAP in reducing CVD risk factors in people with SDB.

DETAILED DESCRIPTION:
It is estimated that 18 million Americans are affected by SDB. SDB involves repeated sleep arousal caused by breathing difficulties. These frequent sleep disruptions may cause a person to experience daytime drowsiness, impaired mental functioning, and trouble concentrating or staying alert. SDB is also associated with an increased risk of certain cardiovascular diseases, such as high blood pressure and heart disease. Researchers believe that increased oxidative stress and inflammation associated with SDB may play a role in the physiologic pathway linking SDB and CVD. However, more information on the SDB-CVD relationship is needed to be able to identify risk factors for CVD and to discover the best means of treatment. CPAP, a current treatment for SDB, acts by delivering air through a mask during sleep. CPAP helps improve overnight breathing and quality of sleep and may, in turn, decrease oxidative stress and associated CVD risks. This study will compare the effectiveness of CPAP versus placebo CPAP in reducing CVD risk factors, such as oxidative stress markers, in people with SDB.

Participation in this study will last between 2.5 and 4 months and will include four to five study visits. During the first study visit, participants will undergo a CPAP titration study, which will involve appropriate CPAP mask fitting and an overnight sleep test to determine the best CPAP pressure, as well as a lower placebo pressure, for each participant. Participants will also be provided educational information on diet, sleep, and the use of CPAP as a treatment for sleep apnea. After the titration study, participants will be asked to wear their fitted CPAP mask every night for the next 2 weeks, during which they will use the lower (placebo) pressure one week and use the higher pressure the other week. During this time, a technician will contact participants every 3 to 4 days to address any questions or problems with the CPAP equipment.

One month later, participants who were able to tolerate and use CPAP most nights will attend Visit 2. This second visit will include an overnight sleep study without wearing the CPAP mask; blood and saliva collection; cheek brushing for genetic material; tests on diabetes, artery stiffness, and circulation; body fat measurements; and questionnaires. Participants will then be randomly assigned to use either the higher pressure CPAP or the lower pressure CPAP for 8 weeks. Visit 3 will occur 1 week after beginning CPAP treatment and will include a fasting blood test. During treatment, participants will be periodically contacted by a technician to check on equipment status.

Upon completing treatment, participants will undergo repeat tests from Visit 2, except that they will wear the CPAP mask in the overnight sleep test. This fourth study visit will mark the completion of treatment for participants assigned to the lower pressure CPAP. Participants assigned to the higher pressure CPAP will be asked to use CPAP for 4 more weeks. These participants will return at the end of the 4 weeks for a final visit, which will include a repeat sleep study and other testing.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe sleep disordered breathing (SDB) (Apnea Hypopnea Index [AHI] greater than or equal to 15) diagnosed within the 2 months before study entry
* Able to participate in more than two overnight/daytime sleep and physiologic assessments over a 2.5-month period

Exclusion Criteria:

* Current or planned use of specific sleep apnea treatments (e.g., CPAP, oral appliance) outside of the study
* Anticipated upper airway surgery or gastric bypass surgery in the 4 months after study completion
* Supplemental oxygen use
* Primary sleep disorder other than sleep apnea (e.g., periodic limb movement disorder)
* Severe chronic insomnia or circadian rhythm disorder with less than 4 hours of sleep per night, chronic problems falling asleep within 1 hour of bedtime, or chronic problems with early morning awakenings
* Unstable medical conditions (e.g., new onset or changing angina; heart attack or congestive heart failure exacerbation documented within the 6 months before study entry; high grade cardiac dysrhythmia/heart block; known unaddressed coronary artery disease by history, angina, stroke, or uncontrolled hypertension or diabetes mellitus; thyroid disorder; cirrhosis; a non-skin cancer diagnosed within the 2 years before study entry)
* Inadequately treated psychiatric disorders or compromised competence
* Daytime sleepiness with reports of sleepiness while driving or during other situations that would present a risk for the subject or public (e.g., operating heavy equipment)
* Alcohol abuse
* Pregnancy
* Use of oral corticosteroids

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2006-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reena Mehra, MD, MS, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mehra R, Storfer-Isser A, Kirchner HL, Johnson N, Jenny N, Tracy RP, Redline S. Soluble interleukin 6 receptor: A novel marker of moderate to severe sleep-related breathing disorder. Arch Intern Med. 2006 Sep 18;166(16):1725-31. doi: 10.1001/archinte.166.16.1725. PMID 16983050
- [Background] Mehra R, Principe-Rodriguez K, Kirchner HL, Strohl KP. Sleep apnea in acute coronary syndrome: high prevalence but low impact on 6-month outcome. Sleep Med. 2006 Sep;7(6):521-8. doi: 10.1016/j.sleep.2006.03.012. Epub 2006 Aug 23. PMID 16931151
- [Background] Mehra R, Benjamin EJ, Shahar E, Gottlieb DJ, Nawabit R, Kirchner HL, Sahadevan J, Redline S; Sleep Heart Health Study. Association of nocturnal arrhythmias with sleep-disordered breathing: The Sleep Heart Health Study. Am J Respir Crit Care Med. 2006 Apr 15;173(8):910-6. doi: 10.1164/rccm.200509-1442OC. Epub 2006 Jan 19. PMID 16424443
- [Derived] May AM, Wang L, Strohl KP, Walia H, Hazen SL, Mehra R. Sex-Specific Differential Responses of Circulating Biomarkers in Obstructive Sleep Apnea Treatment. A Post Hoc Analysis of a Randomized Controlled Trial. Ann Am Thorac Soc. 2020 May;17(5):605-613. doi: 10.1513/AnnalsATS.201908-593OC. PMID 31860326
- [Derived] May AM, Gharibeh T, Wang L, Hurley A, Walia H, Strohl KP, Mehra R. CPAP Adherence Predictors in a Randomized Trial of Moderate-to-Severe OSA Enriched With Women and Minorities. Chest. 2018 Sep;154(3):567-578. doi: 10.1016/j.chest.2018.04.010. Epub 2018 Apr 21. PMID 29684316
- [Derived] DeMartino T, Ghoul RE, Wang L, Bena J, Hazen SL, Tracy R, Patel SR, Auckley D, Mehra R. Oxidative Stress and Inflammation Differentially Elevated in Objective Versus Habitual Subjective Reduced Sleep Duration in Obstructive Sleep Apnea. Sleep. 2016 Jul 1;39(7):1361-9. doi: 10.5665/sleep.5964. PMID 27091532
- [Derived] Paz Y Mar HL, Hazen SL, Tracy RP, Strohl KP, Auckley D, Bena J, Wang L, Walia HK, Patel SR, Mehra R. Effect of Continuous Positive Airway Pressure on Cardiovascular Biomarkers: The Sleep Apnea Stress Randomized Controlled Trial. Chest. 2016 Jul;150(1):80-90. doi: 10.1016/j.chest.2016.03.002. Epub 2016 Mar 18. PMID 26997243

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham CPAP: Participants will receive sham continuous positive airway pressure for a 2 month period. Sham CPAP involves wearing a device that appears similar to a standard CPAP device, but administers a negligible pressure. Adherence will be tracked while the participant wears the device.
  Sham treatment: Participants will use the lower pressure CPAP every night for 8 weeks.
Period: Overall Study
Arm/Group | Sham CPAP | Treatment CPAP
Started (Underwent Randomization) | 77 | 76
Completed Baseline Visit (Completed Baseline Visit) | 74 | 75
Completed 8 Week Visit (Completed 8 Week Visit) | 71 | 72
Completed 12 Week Visit | 0 (12 Week Visit only offered to participants on actual CPAP Treatment) | 29 (12 Week Visit only offered to participants on actual CPAP Treatment)
Completed | 71 | 72
Not Completed | 6 | 4
Not completed — Lost to Follow-up | 4 | 0
Not completed — withdrew due to loss of interest | 0 | 1
Not completed — Withdrew due to osteomyelitis surgery | 0 | 1
Not completed — withdrew could not tolerate CPAP | 0 | 1
Not completed — Declined to be treated | 1 | 0
Not completed — Withdrew due to hypertensive urgency | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment CPAP: Participants will use the higher pressure CPAP, as determined by an in-laboratory attended titration study, every night for 12 weeks.
- Sham CPAP: Participants used the Sham CPAP every night for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Treatment CPAP | Sham CPAP | Total
Number analyzed (Participants) | 75 | 74 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (11.7) | 51.7 (11.8) | 51.0 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 35 | 69
  Male | 41 | 39 | 80
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 37 | 41 | 78
  African American | 36 | 31 | 67
  Other | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 75 | 74 | 149

OUTCOME MEASURES:

1. Primary Outcome: F2-isoprostanes/Cr
Description: Oxidative stress outcome, analyzed absolute change from baseline, with adjustment of baseline
Time Frame: Measured between baseline and after treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/mg
Arm/Group | Sham CPAP | Treatment CPAP
Number analyzed (Participants) | 71 | 72
ng/mg | -0.02 [-0.12 to 0.10] | -0.08 [-0.18 to 0.03]
Statistical Analysis 1: Comparison: Sham CPAP vs Treatment CPAP; Test type: Other; p = 0.38, Regression, Linear; Mean Difference (Final Values) = 0.071, 95% CI 2-sided [-0.090 to 0.23] — F2-isoprostanes/Cr was log-transformed before analysis. The estimation parameter shows the log-transformed mean difference of the absolute change between groups, while the least square means of two groups are transformed back for presentation

2. Primary Outcome: Myeloperoxidase
Description: Oxidative stress outcome, analyzed absolute change from baseline, with adjustment of baseline
Time Frame: Measured between baseline and after treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: pmol/L
Arm/Group | Sham CPAP | Treatment CPAP
Number analyzed (Participants) | 71 | 72
pmol/L | -3.33 [-17.02 to 10.37] | -5.15 [-18.65 to 8.35]
Statistical Analysis 1: Comparison: Sham CPAP vs Treatment CPAP; Test type: Other; p = 0.85, Regression, Linear; Mean Difference (Final Values) = 1.83, 95% CI 2-sided [-17.42 to 21.07]

3. Secondary Outcome: Mean Arterial BP, Evening
Description: Blood pressure outcome, analyzed absolute change from baseline, with adjustment of baseline
Time Frame: Measured between baseline and after treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Sham CPAP | Treatment CPAP
Number analyzed (Participants) | 71 | 72
mm Hg | -0.59 [-2.53 to 1.35] | -0.72 [-2.65 to 1.20]
Statistical Analysis 1: Comparison: Sham CPAP vs Treatment CPAP; Test type: Other; p = 0.92, Regression, Linear; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-2.60 to 2.87]

4. Secondary Outcome: Pulse Wave Velocity, Evening
Description: Pulse wave analysis outcome, analyzed absolute change from baseline, with adjustment of baseline
Time Frame: Measured between baseline and after treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: cm/s
Arm/Group | Sham CPAP | Treatment CPAP
Number analyzed (Participants) | 71 | 72
cm/s | -0.08 [-0.57 to 0.40] | -0.30 [-0.80 to 0.20]
Statistical Analysis 1: Comparison: Sham CPAP vs Treatment CPAP; Test type: Other; p = 0.55, Regression, Linear; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [-0.48 to 0.91]

5. Secondary Outcome: IL-6
Description: Measures of inflammation outcome, analyzed absolute change from baseline, with adjustment of baseline
Time Frame: Measured between baseline and after treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Sham CPAP | Treatment CPAP
Number analyzed (Participants) | 71 | 72
pg/mL | 0.29 [-0.10 to 0.68] | -0.08 [-0.46 to 0.29]
Statistical Analysis 1: Comparison: Sham CPAP vs Treatment CPAP; Test type: Other; p = 0.17, Regression, Linear; Mean Difference (Final Values) = 0.38, 95% CI 2-sided [-0.16 to 0.92]

6. Secondary Outcome: Mean Arterial BP, Morning
Description: Blood pressure outcome, analyzed absolute change from baseline, with adjustment of baseline
Time Frame: Measured between baseline and after treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Sham CPAP | Treatment CPAP
Number analyzed (Participants) | 71 | 72
mm Hg | 0.24 [-1.64 to 2.12] | -2.17 [-4.03 to -0.30]
Statistical Analysis 1: Comparison: Sham CPAP vs Treatment CPAP; Test type: Other; p = 0.076, Regression, Linear; Mean Difference (Final Values) = 2.40, 95% CI 2-sided [-0.26 to 5.07]

7. Secondary Outcome: sIL-6R
Description: Measures of inflammation outcome, logarithm transformed before analysis due to skewed distribution, analyzed change of from baseline with adjustment of baseline. The least squares mean is transformed back to present the percent change from baseline.
Time Frame: Measured between baseline and after treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Sham CPAP | Treatment CPAP
Number analyzed (Participants) | 71 | 72
percent change | 0.02 [-0.02 to 0.06] | -0.04 [-0.08 to -0.01]
Statistical Analysis 1: Comparison: Sham CPAP vs Treatment CPAP; Test type: Other; p = 0.019, Regression, Linear; Mean Difference (Final Values) = 0.062, 95% CI 2-sided [0.010 to 0.11] — sIL-6R was log-transformed before analysis. The estimation parameter shows the log-transformed mean difference of the absolute change between groups, while the least square means of two groups are transformed back for presentation

8. Secondary Outcome: Pulse Wave Velocity, Morning
Description: Pulse wave analysis outcome, analyzed absolute change from baseline, with adjustment of baseline
Time Frame: Measured between Months 2 and 3 of treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: cm/s
Arm/Group | Sham CPAP | Treatment CPAP
Number analyzed (Participants) | 71 | 72
cm/s | -0.25 [-0.82 to 0.32] | -0.42 [-1.01 to 0.16]
Statistical Analysis 1: Comparison: Sham CPAP vs Treatment CPAP; Test type: Other; p = 0.68, Regression, Linear; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [-0.64 to 0.99]

9. Secondary Outcome: Augmentation Index, Evening
Description: Pulse wave analysis outcome (a ratio of the augmentation of central aortic pressure by a reflected pulse wave, calculated from the blood pressure waveform), analyzed absolute change from baseline, with adjustment of baseline
Time Frame: Measured between Months 2 and 3 of treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Sham CPAP | Treatment CPAP
Number analyzed (Participants) | 71 | 72
percent change | -0.43 [-3.87 to 3.00] | -1.79 [-5.36 to 1.78]
Statistical Analysis 1: Comparison: Sham CPAP vs Treatment CPAP; Test type: Other; p = 0.59, Regression, Linear; Mean Difference (Final Values) = 1.35, 95% CI 2-sided [-3.60 to 6.31]

10. Secondary Outcome: Augmentation Index, Morning
Description: as for outcome 9
Time Frame: Measured between Months 2 and 3 of treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Sham CPAP | Treatment CPAP
Number analyzed (Participants) | 71 | 72
percent change | 0.44 [-2.22 to 3.10] | -6.49 [-9.32 to -3.65]
Statistical Analysis 1: Comparison: Sham CPAP vs Treatment CPAP; Test type: Other; p < 0.001, Regression, Linear; Mean Difference (Final Values) = 6.93, 95% CI 2-sided [3.04 to 10.81]

ADVERSE EVENTS:
Groups:
- SHAM CPAP: Participants will receive sham continuous positive airway pressure for a 2 month period. Sham CPAP involves wearing a device that appears similar to a standard CPAP device, but administers a negligible pressure. Adherence will be tracked while the participant wears the device.
  Sham CPAP: Participants will use the lower pressure CPAP every night for 8 weeks.
- Run-in/Washout Treatment CPAP: The initial run-in and washout period for study qualification to document CPAP adherence on treatment CPAP.
- Run-in/Washout Sham CPAP: The initial run-in and washout period for study qualification to document CPAP adherence on Sham CPAP (negligible pressure).
Arm/Group | SHAM CPAP | Treatment CPAP | Run-in/Washout Treatment CPAP | Run-in/Washout Sham CPAP
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/76 | 0/153 | 0/153
Serious Adverse Events (participants affected / at risk) | 3/77 | 3/76 | 6/153 | 2/153
Other Adverse Events (participants affected / at risk) | 27/77 | 32/76 | 23/153 | 8/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SHAM CPAP (N=77) | Treatment CPAP (N=76) | Run-in/Washout Treatment CPAP (N=153) | Run-in/Washout Sham CPAP (N=153)
Chest Pain (went to ER) (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Enlarged coronary artieries/chest pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irregular heartbeat (went to ER) (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
New onset atrial flutter (shown on psg) (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ER with swollen Knee (hospitalized) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hospitalized for seizures (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration and possible kidney failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia/Influenza (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Spot on lung - biopsy for cancer (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foot ulcer amputation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ruptured appendix (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SHAM CPAP (N=77) | Treatment CPAP (N=76) | Run-in/Washout Treatment CPAP (N=153) | Run-in/Washout Sham CPAP (N=153)
Bruise from venipucture (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nose bleeding (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Elevated blood pressure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heart monitor for irregular heartbeat (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Run of nonsustained ventricular tachycardia on PSG (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cataract surgery (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye infection/injury (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal cramping (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Elevated glucose level (Metabolism and nutrition disorders) | 13 (13) | 11 (11) | 0 (0) | 0 (0)
Chronic pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Developed sciatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fell and bruised rib (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General pain (leg, back, muscle) (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Hand injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Knee replacement (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
auto accident / physical therapy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headaches (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Breathing problems (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cold/congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 4 (4) | 0 (0)
Dry cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-productive cough/post nasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus infection (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 2 (2) | 2 (2)
Spot on lung (possible cancer) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Strep throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abrasion on bridge of nose from CPAP mask (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cysts on chin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flare up of eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Redness on external nares from nasal pillow mask marks on face from maks (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tumor removed from finger (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ulcer on foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
scabs on head from electrodes from psg (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Kidney Stone (Surgical and medical procedures) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Tooth extracted/root canal (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes